CLINICAL TRIAL: NCT03513705
Title: Impact of Nationwide Enhanced Implementation of Best Practices in Pancreatic Cancer Care (PACAP-1): a Multicenter Stepped-wedge Cluster Randomized Controlled Trial
Brief Title: Impact of Nationwide Enhanced Implementation of Best Practices in Pancreatic Cancer Care (PACAP-1)
Acronym: PACAP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Cancer Society (Other); Comprehensive Cancer Centre The Netherlands (Other)
Responsible Party: Principal Investigator, M.G. Besselink, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: W17_454; UVA 2013-5842 (Other Grant/Funding Number: Alpe d'HuZes / Dutch Cancer Society (KWF))
Record Dates: First submitted 2018-04-12; First posted 2018-05-01 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: implementation; randomized trial; pancreatic cancer; nationwide; survival; quality of life
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best practice (Experimental): Enhanced implementation of best practices in pancreatic cancer care
  Interventions: Other: Best practices in pancreatic cancer care
- Current practice (No Intervention): Pancreatic cancer care according to current practice

INTERVENTIONS:
Other: Best practices in pancreatic cancer care — All best practices follow the current state of the Dutch guideline on pancreatic cancer and the literature.
  Arms: Best practice

SUMMARY:
PACAP-1 will evaluate to what extent an enhanced implementation of best practices in pancreatic cancer care leads to a prolonged survival and improvement of quality of life as compared to current practice.

DETAILED DESCRIPTION:
Rationale:

The Dutch Pancreatic Cancer Project (PACAP) is an initiative of the Dutch Pancreatic Cancer Group and was officially launched in July 2014. PACAP is 1 of the largest nationwide collaborative outcomes registration and biobanking projects on pancreatic and periampullary cancer worldwide and includes the Dutch Pancreatic Cancer Audit (DPCA), the Patient Reported Outcome Measures (PROMs), an online expert panel, and the Netherlands Cancer Registry (NCR, Netherlands Comprehensive Cancer Organization; IKNL). During the first 3 years of PACAP, regional variations in treatment and guideline (non-)compliance were observed. These differences may lead to differences in survival and quality of life of pancreatic cancer patients throughout the Netherlands. From PACAP data and literature, best practices for pancreatic cancer care have been identified.

Objective:

The aim of PACAP-1 is to evaluate to what extent an enhanced implementation of best practices in pancreatic cancer care in the Netherlands leads to a prolonged survival and improvement of quality of life as compared to current practice.

Study design:

The PACAP-1 trial is a nationwide stepped-wedge cluster randomized controlled trial. In a per center stepwise and randomized manner, best practices in pancreatic cancer care are implemented in all 17 Dutch pancreatic centers. A regional pancreatic cancer team will be established per pancreatic center that functions as point of contact for peripheral centers in the region. Patient outcomes and compliance will be monitored by the registries founded in the PACAP initiative.

Study Population:

Prospective cohort of all pancreatic cancer patients diagnosed and treated in the Netherlands.

Interventions:

Best practices will be implemented in 3 key medical specialties in pancreatic cancer care: medical oncology, surgery and gastroenterology. Best practices will be implemented in centers during a 6 week intensive initiation period which includes monitoring, return visits, provider feedback in combination with education and reminders. The best practices follow the Dutch guideline on pancreatic cancer and the current state of the literature and can be executed without additional overall costs per center.

Main study outcomes:

The primary outcome is 1-year overall survival. Secondary outcomes include quality of life (first secondary outcome), 3- and 5-year overall survival and success of implementation of every PACAP-1 intervention and participation in DPCG randomized trials.

ELIGIBILITY:
Inclusion Criteria patients:

* All pancreatic cancer patients

Exclusion Criteria patients:

* There are no specific exclusion criteria

Inclusion Criteria clusters:

* All 17 centers of the DPCG. These centers each perform >20 pancreatoduodenectomies (PDs) annually. Each center already has a coordinating role for pancreatic cancer for its region. It is expected that the enhanced implementation of best practices will have an impact in the entire local network

Exclusion Criteria clusters:

* There are no specific center exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
1-year overall survival | 1-year
  Overall survival 1-year after diagnosis of pancreatic cancer

SECONDARY OUTCOMES:
3-year overall survival | 3-year
  Overall survival 3-year after diagnosis of pancreatic cancer
5-year overall survival | 5-year
  Overall survival 5-year after diagnosis of pancreatic cancer
Complications | Through study completion, on average up to 25 months
  Complications of chemotherapy (toxicity grade 3-4 and type of toxicity) and biliary stent placement
Effect of implementation of best practices | Through study completion, on average up to 25 months
  Proportion of patients that underwent the separate best practice interventions if applicable
Registry outcomes | Through study completion, on average up to 25 months
  Best practice registrations measured through Patient Reported Outcome Measures
Registry outcomes | Through study completion, on average up to 25 months
  Best practice registrations measured through the Dutch Pancreatic Cancer Audit
Registry outcomes | Through study completion, on average up to 25 months
  Best practice registrations measured through the Netherlands Cancer Registry
Use of smartphone application | Through study completion, on average up to 25 months

OTHER OUTCOMES:
Quality of life with Area Under the Curve (AUC) up to 1 year after diagnosis | up to 1 year after diagnosis
  Quality of life with Area Under the Curve (AUC) up to 1 year after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Marc Besselink, Prof. Dr., Principal Investigator — Academic Medical Center - Cancer Center Amsterdam
Locations (17):
- Netherlands (17):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Academic Medical Center, Amsterdam
  - Onze Lieve Vrouwen Gasthuis, Amsterdam
  - VU Medical Center, Amsterdam
  - Amphia, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Catharina, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Tjongerschans, Heerenveen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - RAKU (University Medical Center Utrecht and Sint Antonius Ziekenhuis), Utrecht
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
De-identified data generated during the PACAP-1 trial will be made available to other researcher upon request from Marc Besselink and/or the Dutch Pancreatic Cancer Group (DPCG)
Supporting Information: Study Protocol
Time Frame: Upon request
Access Criteria: Upon request
URL: http://www.dpcg.nl

REFERENCES:
- [Derived] Seelen LWF, Augustinus S, Stoop TF, Bouwense SAW, Busch OR, Cirkel GA, van Eijck CHJ, de Vos-Geelen J, Groot Koerkamp B, Haj Mohammad N, de Hingh IHJT, van Alphen E, Homs MYV, Liem MSL, Los M, de Meijer VE, Mekenkamp LJM, Sprangers MAG, Stommel MWJ, Wilmink JW, Besselink MG, van Santvoort HC, van Laarhoven HWM, Molenaar IQ; Dutch Pancreatic Cancer Group. Quality of Life Among Patients With Locally Advanced Pancreatic Cancer: A Prospective Nationwide Multicenter Study. J Natl Compr Canc Netw. 2025 Feb 19;23(3):97-104. doi: 10.6004/jnccn.2024.7091. PMID 39970867
- [Derived] Mackay TM, Latenstein AEJ, Augustinus S, van der Geest LG, Bogte A, Bonsing BA, Cirkel GA, Hol L, Busch OR, den Dulk M, van Driel LMJW, Festen S, de Groot DA, de Groot JB, Groot Koerkamp B, Haj Mohammad N, Haver JT, van der Harst E, de Hingh IH, Homs MYV, Los M, Luelmo SAC, de Meijer VE, Mekenkamp L, Molenaar IQ, Patijn GA, Quispel R, Romkens TEH, van Santvoort HC, Stommel MWJ, Venneman NG, Verdonk RC, van Vilsteren FGI, de Vos-Geelen J, van Werkhoven CH, van Hooft JE, van Eijck CHJ, Wilmink JW, van Laarhoven HWM, Besselink MG; Dutch Pancreatic Cancer Group. Implementation of Best Practices in Pancreatic Cancer Care in the Netherlands: A Stepped-Wedge Randomized Clinical Trial. JAMA Surg. 2024 Apr 1;159(4):429-437. doi: 10.1001/jamasurg.2023.7872. PMID 38353966
- [Derived] Mackay TM, Smits FJ, Latenstein AEJ, Bogte A, Bonsing BA, Bos H, Bosscha K, Brosens LAA, Hol L, Busch ORC, Creemers GJ, Curvers WL, den Dulk M, van Dieren S, van Driel LMJW, Festen S, van Geenen EJM, van der Geest LG, de Groot DJA, de Groot JWB, Haj Mohammad N, Haberkorn BCM, Haver JT, van der Harst E, Hemmink GJM, de Hingh IH, Hoge C, Homs MYV, van Huijgevoort NC, Jacobs MAJM, Kerver ED, Liem MSL, Los M, Lubbinge H, Luelmo SAC, de Meijer VE, Mekenkamp L, Molenaar IQ, van Oijen MGH, Patijn GA, Quispel R, van Rijssen LB, Romkens TEH, van Santvoort HC, Schreinemakers JMJ, Schut H, Seerden T, Stommel MWJ, Ten Tije AJ, Venneman NG, Verdonk RC, Verheij J, van Vilsteren FGI, de Vos-Geelen J, Vulink A, Wientjes C, Wit F, Wessels FJ, Zonderhuis B, van Werkhoven CH, van Hooft JE, van Eijck CHJ, Wilmink JW, van Laarhoven HWM, Besselink MG; Dutch Pancreatic Cancer Group. Impact of nationwide enhanced implementation of best practices in pancreatic cancer care (PACAP-1): a multicenter stepped-wedge cluster randomized controlled trial. Trials. 2020 Apr 16;21(1):334. doi: 10.1186/s13063-020-4180-z. PMID 32299515